CLINICAL TRIAL: NCT04691752
Title: Management of Patients With Chronic Obstructive Pulmonary Disease in Granada: a Clinical Audit
Acronym: Epocap
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Andalusian School of Public Health (Other Government)
Collaborators: Hospital de Alta Resolución de Loja. Agencia Sanitaria Hospital de Poniente (Unknown)
Responsible Party: Sponsor
Other Study IDs: EASP-EPOC-18
Record Dates: First submitted 2020-12-17; First posted 2020-12-31 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: COPD
Keywords: COPD; Emphysema; Chronic Bronchitis; Clinical audit; Primary Healthcare
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients: * Adults (men or women) aged more than 40 years old
  * Diagnostic code in Andalusian clinical records (Diraya) in accordance with ICD-9 (Diagnostic codes 496, 492.8, 494.0, 491.20, 493.2)
  * Current of former smokers of at least 10 pack- years
  * Patient with a minimum follow up of 1 year, who have been assisted in a scheduled primary care appointment at inclusion date.
  Interventions: Other: Audit

INTERVENTIONS:
Other: Audit — Audit from clinical records

SUMMARY:
It is actually unknown how are the COPD clinical guidelines followed in primary care in Andalusia, specially for diagnosis and follow up of patients with this diseases. Detection of areas for improvement in COPD healthcare can be useful in order to implement improvement programs. This project is a clinical audit among primary care centres in Granada attending patients with COPD in the public health system

DETAILED DESCRIPTION:
The aim of this study is to audit the attention to people with COPD among primary care centres in Granada, as well as how clinical guidelines are followed and other recommendations. The study will comprise medical records from more than 3000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (men or women) aged more than 40 years old
* Diagnostic code in Andalusian clinical records (Diraya) in accordance with ICD-9 (Diagnostic codes 496, 492.8, 494.0, 491.20, 493.2)
* Current of former smokers of at least 10 pack- years
* Patient with a minimum follow up of 1 year, who have been assisted in a scheduled primary care appointment at inclusion date.

Exclusion Criteria:

* Patients with a diagnostic code for COPD attended at primary care office, but without information related with COPD in the previous year.
* Patients currently involved in any clinical trial or research study related with COPD.
* Those patients excluded will be collected in an exclusion causes chart for each centre. These patients will not affect overall number of patients targeted for each centre.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnostic code for COPD in Andalusian health records- Diraya-(ICD 9 Diagnostic codes 496, 492.8, 494.0, 491.20, 493.2)attended for any reason in a scheduled primary care office in Granada. Selection process of participant centres will be performed aiming to reflect proportionally the population distribution of Granada province and certain circumstances such as population density of some of the counties
Sampling Method: Non-Probability Sample
Enrollment: 2280 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
To audit public healthcare for patients with COPD in primary care offices in Granada. | 1 year
  Number of patients with a diagnosis code for COPD among participants with auitable clinical records

SECONDARY OUTCOMES:
To describe clinical profile of patients with COPD attended at primary care offices in Granada | 1 year
  Number of patients auditable with a diagnosis code for COPD attended at primary care center
To describe the quality of care for COPD patients, focusing on determinants of variability(such as seasonality) | 1 year
  Pproportion of patients receiving correct diagnosis for COPD based on spirometric measurements
To evaluate the adherence to clinical guidelines for COPD | 1 year
  Proportion of patients with COPD with correct diagnosis according to GesEPOC guidelines.
To describe current available resources for COPD healthcare in the primary care level in Granada. | 1 year
  Number of centers with spirometry available

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request
Supporting Information: Study Protocol, CSR
Time Frame: When recruitment is finished